CLINICAL TRIAL: NCT07253545
Title: IOBBAT - Impact of Basic Body Awareness Therapy on Body Awareness
Acronym: IOBBAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Medical University of Graz (Other); FH Joanneum Gesellschaft mbH (Industry); Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IOBBAT_1
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Perception, Self; Body Awareness; Self-Assessment
Keywords: Basic Body Awareness Therapy; Body awareness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Body Awareness Therapy (Active Comparator): Basic Body Awareness Therapy (BBAT) is a treatment method that uses the body and its movements as a foundation for improved health. It incorporates everyday movements, Western therapeutic techniques, and elements from Tai Chi to enhance balance, stability, and movement quality. The exercises are simple to perform and focus attention on postural control and stability, breathing, and mental presence. The goal is to strengthen the individual's health resources, thereby promoting autonomy, activity, and participation.
  Interventions: Procedure: Basic Body Awareness Therapy
- Lecture (Placebo Comparator): The control group receives a 20-minute video-based lecture on medicinal herbs
  Interventions: Other: Lecture

INTERVENTIONS:
Procedure: Basic Body Awareness Therapy — Basic Body Awareness Therapy (BBAT) is a treatment method that uses the body and its movements as a foundation for improved health. It incorporates everyday movements, Western therapeutic techniques, and elements from Tai Chi to enhance balance, stability, and movement quality. The exercises are simple to perform and focus attention on postural control and stability, breathing, and mental presence. The goal is to strengthen the individual's health resources, thereby promoting autonomy, activity, and participation.
  Arms: Basic Body Awareness Therapy
Other: Lecture — The control group receives a 20-minute video-based lecture on medicinal herbs
  Arms: Lecture

SUMMARY:
Body awareness (BA) is an essential factor for health and well-being. In 2021, the IOBA (Impact on Body Awareness) study was conducted at the Institute of Physical Medicine & Rehabilitation at Kepler University Hospital (Clinical Trials NCT05004272). This study investigated the effects of massage and gymnastics on BA in healthy individuals. The protocol provides a solid foundation for further research projects on BA. The aim of the present study is to examine the immediate effects of a Basic Body Awareness Therapy (BBAT) session compared to a lecture (control group) on BA and well-being, and to explore correlations with BA.

In a randomized controlled study with 60 physiotherapy students in two groups (BBAT and control group) the use of the ABC questionnaire and further German questionnaires (Short questionnaire on self-perception of the body, self-rating mood scale - revised) concerning body awareness and well-being should analyse the following hypothesis: There is a difference in the change of BA between intervention (BBAT) and control group, Before interventions demographic data and further questionnaires concerning health conditions of the participants (e.g. Simple Physical Activity Questionnaire, Short Form Health Survey, Brief Symptom Inventory) are administered. Correlations between BA and the results of these tests will be investigated too. All these analyses can provide insights into the effects of BBAT on BA. The identification of patterns in BA among students can be used for future comparisons with patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Students in the 5th semester of the Bachelor's degree program in physiotherapy at FH JOANNEUM in Graz
* Signed informed consent for participation

Exclusion Criteria:

* Pregnancy
* Current illnesses or injuries that represent a contraindication for participating in the BBAT session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Awareness Body Chart Questionnaire | Before intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness. In the case of pain, the pain location can also be marked on the body chart with a red pen and recorded on a 100 mm Visual Analogue Scale from 0 (no pain) to 100 (unbearable pain).
Awareness Body Chart Questionnaire | Immediately after intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness. In the case of pain, the pain location can also be marked on the body chart with a red pen and recorded on a 100 mm Visual Analogue Scale from 0 (no pain) to 100 (unbearable pain).

SECONDARY OUTCOMES:
Short questionnaire on self-perception of the body | Before intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Short questionnaire on self-perception of the body | Immediately after intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Self-rating mood scale - revised | Before intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.
Self-rating mood scale - revised | Immediately after intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.

OTHER OUTCOMES:
Simple Physical Activity Questionnaire | Before intervention
  Questionnaire to survey physical activity: It should show a snapshot of hours per day of an average day in the past week. The time in bed, the time while doing sedentary work (including dozing), while walking, while exercising and during other physical activities (such as household chores) is interrogated. The test does not measure the intensity of physical activity, but rather sorts it into the groups walking, sport and other categories.
Short Form Health Survey (SF-12) | Before intervention
  Questionnaire on health-related quality of life. It consists of twelve questions relating to the last four weeks and yields statements about eight different dimensions of subjective health: general health perception, physical health, physically-conditioned role function, physical pain, vitality, mental health, emotionally-related role function, social functionality. Different Likert-Scales are used. A physical sum scale and a psychological sum scale can be calculated. The polarity of four items must be reversed so that higher values in all items and total scales reflect a better state of health. Normative data are available.
Brief Symptom Inventory (BSI) | Before intervention
  Questionnaire on the burden of symptoms. The BSI is also called the Brief Symptom Check List (BSCL), it is a short form of the SCL-90 (Derogatis, 1993). The BSI consists of 53 items (physical as well as psychological symptoms), which are assessed subjectively on a Likert scale in relation to the last seven days from 0 = "not at all" to 5 = "very strong". The items result in nine scales: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.
Beck Depression Inventory II (BDI-II) | Before intervention
  The BDI-II represents a self-rating instrument to assess the severity of depression. Four statements are given for each of 21 questions, from which the one that best describes how the person has felt in the past week is to be selected. In scoring, each item is given a score of 0 to 3, depending on the choice (higher number means higher depression scores), and after directly adding the scores of the individual items, a total score of 0 to 63 is obtained.
Insomnia Severity Index (ISI) | Before intervention
  The ISI is a self-assessment questionnaire used to evaluate the nature, severity, and impact of insomnia over the past two weeks. The ISI contains seven items rated with a five-point Likert scale (0 = not at all, 4 = very severe problem), with the total score ranging from 0 to 28. Higher scores indicate greater severity of insomnia. Scores from 0-7 are considered no insomnia, 8-14 is subthreshold insomnia, 15-21 is moderate insomnia, and 22-28 is severe insomnia.
Body Mass Index | Before intervention
  Relation of body weight to the square of body height
Like/Dislike Body Chart | Before intervention
  As an extension to the ABC, this questionnaire is intended to answer the question of whether there are areas of the body that one particularly likes about oneself or that one dislikes about oneself. If yes, one can draw these with a purple color pencil ("particularly like") and/or with a gray color pencil ("do not like") in an extra Body Chart.
Additional questions | Before intervention
  Questions on demographic data and chronic complaints and current illnesses

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mittermaier, M.D., Study Director — Kepler University Clinic, Dept. of Physical Medicine & Rehabilitation

IPD SHARING:
Plan to Share IPD: No